CLINICAL TRIAL: NCT03404414
Title: Detection of Functioning Pituitary Microadenoma With Inconclusive MRI Findings: PET/MRI Versus PET/CT
Brief Title: Detection of Functioning Pituitary Microadenoma: PET/MRI Versus PET/CT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NM017
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FDG PET/MRI and 18F-FDG PET/CT (Experimental): The patients were injected with 370 MBq of 18F-FDG in one dose intravenously and underwent PET/MRI or PET/CT scan 1 hour later
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — Single-dose 18F-FDG were injected into the patients before the PET/MR or PET/CT scans.
  patients before the PET/CT scans

SUMMARY:
This is a prospective case-control study to compare the usefulness of 18F-FDG PET/MRI with that of 18F-FDG PET/CT in detection of functioning pituitary microadenomas.A single dose of 370 Mega-Becquerel (MBq) 18F-FDG will be injected intravenously.Visual and semiquantitative method will be used to assess the PET/MRI and PET/CT images.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) may be insufficient to locate functioning pituitary microadenoma.This study compared the usefulness of 18F-FDG PET/MRI with that of 18F-FDG PET/CT in detection of functioning pituitary microadenomas in patients with inconclusive conventional MRI findings. Trans-sphenoidal adenomectomy was performed within 2 weeks of imaging.The PET/CT and PET/MRI findings and tracer uptake levels were correlated with the surgical findings and pathological results.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were pathologically diagnosed with pituitary adenoma after surgery were recruited, and were able to provide basic information and sign the written informed consent form.

Exclusion Criteria:

* The exclusion criteria included claustrophobia, kidney or liver failure, and inability to fulfill the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 18F-FDG in pituitary adenoma | 5 years
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in pituitary adenoma will be measured

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, M.D.,PhD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China